CLINICAL TRIAL: NCT06063135
Title: Effects of Physical Exercise Timing On Strength and Cardiometabolic Health
Acronym: EPOCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Raphael Knaier, Researcher Group leader: Circadian Exercise, University of Basel
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EPOCH
Record Dates: First submitted 2023-09-18; First posted 2023-10-02 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Physical Inactivity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Single life-style coaching session
- Exercise Time 1 (Experimental): Physical exercise intervention taking place at one time of the day
  Interventions: Other: Physical Exercise Intervention
- Exercise Time 2 (Experimental): Physical exercise intervention taking place at another time of day
  Interventions: Other: Physical Exercise Intervention

INTERVENTIONS:
Other: Physical Exercise Intervention — Two strength training session per week and one endurance training session per week
  Arms: Exercise Time 1; Exercise Time 2

SUMMARY:
Physical exercise is well known to improve human health. Current guidelines provide recommendations on the frequency, intensity, type and duration of exercise. However, they do not provide recommendations for the time of day, exercise should be performed. This is surprising considering that the influence of timing of behaviors such as sleep or nutrition as well as the impact of the circadian timing system on health are well documented. Further, there is evidence for diurnal variation in maximum performance which enables individuals to exercise with different intensities at different times of day, which in the long term might affect physical adaptations to exercise. Thus, this research study investigates if exercise timing impacts human health.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 30 kg/m2

Exclusion Criteria:

* Structured resistance training within the last six months
* Ongoing shift work
* Irregular bedtime (> 2 hours variation in habitual bed time)
* Smoking
* Travels across more than two time zones within the last four weeks
* Inability to follow the study procedures (e.g. due to language barriers, psychological disorders, dementia, etc.)
* Known pregnancy or lactating women
* Participation in any other clinical trial within the last four weeks
* Medical condition that is a contra indicator for resistance training, endurance training, or exercising until maximum exhaustion including insufficiently controlled blood pressure (systolic > 170 mmHg, diastolic > 100 mmHg), ongoing cancer treatment, unstable angina pectoris, uncontrolled bradyarrhythmia or tachyarrhythmia, severe uncorrected valvular heart disease, clinically relevant acute infection, any form of musculoskeletal injury, orthopedic problems or decompensated cardiovascular disease
* Insulin dependent diabetes
* Participants using metformin

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Maximum strength | Pre-Intervention (i.e. 1 to 28 days before the first training session of the exercise intervention) and Post-Intervention (i.e. 1 to 28 days after the last training session of the exercise intervention)
  Mean value of the maximum isometric strength assessed at four different times of the day with an isometric mid-thigh pull on a force plate.

SECONDARY OUTCOMES:
Glucose control | Pre-Intervention (i.e. 1 to 28 days before the first training session of the exercise intervention) and Post-Intervention (i.e. 1 to 28 days after the last training session of the exercise intervention)
  2-h postprandial area under the curve for glucose after an oral glucose tolerance test
Body composition | Pre-Intervention (i.e. 1 to 28 days before the first training session of the exercise intervention) and Post-Intervention (i.e. 1 to 28 days after the last training session of the exercise intervention)
  total body fat mass assessed with DXA
Cardiorespiratory fitness | Pre-Intervention (i.e. 1 to 28 days before the first training session of the exercise intervention) and Post-Intervention (i.e. 1 to 28 days after the last training session of the exercise intervention)
  VO2max assessed with cardiopulmonary exercise test

CONTACTS AND LOCATIONS:
Overall Officials: Raphael Knaier, PhD, Principal Investigator — University of Basel
Locations (1):
- University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be provided in a data repository in accordance to FAIR principles
Time Frame: After completion of study